CLINICAL TRIAL: NCT03531827
Title: A Single Arm Phase II Study Combining CRLX101, a Nanoparticle Camptothecin, With Enzalutamide in Patients With Progressive Metastatic Castration Resistant Prostate Cancer Following Prior Enzalutamide Treatment
Brief Title: Combining CRLX101, a Nanoparticle Camptothecin, With Enzalutamide in People With Progressive Metastatic Castration Resistant Prostate Cancer Following Prior Enzalutamide Treatment
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed for toxicity.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 180096; 18-C-0096
Record Dates: First submitted 2018-05-18; First posted 2018-05-22 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Castration Resistant Prostate Cancer; Prostate Neoplasms
Keywords: Androgen Receptor Antagonist; PSA; Hormonal Therapy; Nanoparticle Drug; Antitumor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; IT-101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Lead-In Safety: CRLX101 with Enzalutamide (Experimental): Combination treatment of increasing dose of CRLX101 (formerly IT-101) with enzalutamide
  Interventions: Drug: enzalutamide; Drug: CRLX101
- 2/Efficacy: CRLX101 with Enzalutamide (Experimental): Tolerable dose of CRLX101 (formerly IT-101) in combination with enzalutamide (8 participants, expandable to 21 total participants)
  Interventions: Drug: enzalutamide; Drug: CRLX101

INTERVENTIONS:
Drug: enzalutamide — enzalutamide is an androgen receptor (AR) antagonist that is standard care therapy for metastatic prostate cancer
  Other Names: Xtandi
Drug: CRLX101 — CRLX101 is a nanoparticle-drug conjugate (NDC) comprised of a linear cyclodextrin-polyethylene glycol-base polymer conjugated to multiple 2 (S)-camptothecin (CPT) molecules (Poly-CD-PEG-Camptothecin)
  Other Names: IT-101

SUMMARY:
Background:

Some prostate cancer keeps growing even when testosterone in the body drops to very low levels. This is called castrate-resistant prostate cancer. One treatment is enzalutamide. This is a modern hormonal therapy. But it only works for a certain amount of time and then the cancer becomes resistant to it. Researchers want to see if adding the treatment CRLX101 (formerly IT-101) could make enzalutamide work again for people who have already had it.

Objective:

To test a new way of treating prostate cancer using CRLX101 plus enzalutamide in people with certain prostate cancer who already had enzalutamide treatment.

Eligibility:

Adults ages 18 years and older with metastatic, castration-resistant prostate cancer who have had enzalutamide treatment

Design:

Participants will be screened with a medical history and physical exam. They will have blood and urine tests. They will have a scan of the chest/abdomen/pelvis. They will have a bone scan.

Participants will get treatment in cycles. A cycle lasts 28 days. They will take enzalutamide by mouth once a day. They will get CRLX101 through an intravenous (IV) every 1 or 2 weeks.

Participants will repeat screening tests throughout the study.

Participants will have a follow-up visit 3-4 weeks after they stop taking the study drug. They will repeat most screening tests and have an electrocardiogram.

DETAILED DESCRIPTION:
Background:

* Enzalutamide is established as first-line hormonal therapy in participants with metastatic castration resistant prostate cancer (mCRPC). However, it is increasingly recognized that acquired resistance to therapy (e.g., androgen receptor (AR) overexpression, androgen receptor variant 7 (AR-V7) could limit the durability of response to therapy
* Upregulation of Hypoxia-inducible factor 1-alpha (HIF-1Alpha) in hypoxic tumor cells provides a mechanism of acquired resistance to current hormonal therapies and chemotherapies. Acquired resistance increases angiogenesis and metastasis, leading to disease progression
* Targeting the hypoxia driven tumor microenvironment (e.g., down-regulation of HIF-1Alpha) in addition to the androgen receptor (e.g., enzalutamide) has synergistic activity against prostate cancer cell line models (e.g., LNCaP, 22Rv1).
* CRLX101 is a nanoparticle drug conjugate composed of 20(S)-camptothecin (a potent and highly selective topoisomerase I inhibitor with anti-HIF-1Alpha properties) conjugated to a linear, cyclodextrin-polyethylene glycol-based polymer
* CRLX101 has been shown to be safe, tolerable, and efficacious in numerous Phase II clinical investigations in a variety of tumor subtypes.
* Preclinical and clinical studies have shown CRLX101 significantly down-regulates HIF-1alpha, impacting tumor-driven angiogenesis.
* The treatment combination of CRLX101 and enzalutamide provides a reasonable approach to re-sensitizing prostate cancer cells to hormonal therapy via synergistic antitumor activity and inhibition of acquired resistance

Objectives:

-Primary Objective: To evaluate the anti-tumor activity of CRLX101 at the recommended phase II dose (RP2D) in combination with enzalutamide with respect to treatment response, defined as greater than or equal to 50% PSA decline or stable disease on imaging following 5 months of treatment.

Eligibility:

* Patients must have progressive mCRPC per Prostate Cancer Working Group 3(PCWG3)
* Patients must be at least 18 years of age and able to give informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2
* Evaluable metastatic disease on bone scan or measurable disease on computed tomography (CT) Scan per PCWG3 and/or Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients must have had disease progression while receiving prior enzalutamide treatment

Design:

* The study will be conducted using an optimal two stage Phase II design (8 participants, expandable to 21 participants total) aimed to determine the percentage of participants with a prostate-specific antigen (PSA) decline of greater than 50% or stable disease at 5 months.
* The first 3 to 6 participants enrolled on study will follow a lead-in dosing scheme to confirm the safety of the combination (CRLX101 12 mg/m(2) every 2 weeks for the first two cycles, followed by CRLX101 15 mg/m(2) every 2 weeks at the start of cycle 3, with enzalutamide 160 mg administered once daily starting on cycle 1 day 2) prior to initiation of the optimal two stage study design.
* For participants enrolled on study following the lead-in, the confirmed tolerable dose of CRLX101 will be administered via intravenous (IV) infusion every 2 weeks. Enzalutamide 160 mg will be administered orally once daily beginning on cycle 1 day 2.
* Blood and urine will be collected at multiple time points for pharmacokinetic (PK) and pharmacodynamic (PD0 analyses.
* Tumor assessments will be made using Technetium-99 (99Tc) bone scintigraphy and/or CT scan (chest, abdomen, and pelvis) at baseline, prior to Cycle 3 and every 3 cycles thereafter.
* The accrual ceiling for the study is set at 30 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed prostate cancer confirmed by either the Laboratory of Pathology at the national Institutes of Health (NIH) Clinical Center or Walter Reed National Military Medical Center at Bethesda prior to starting this study. If no pathological specimen is available, patients may enroll with a pathologist's report showing a histological diagnosis of prostate cancer and clinical course consistent with the disease.
* Patients must have progressive metastatic castration-resistant prostate cancer mCRPC. There must be radiographic evidence of disease progression or biochemically (rising prostate-specific antigen (PSA) levels on successive measurements) recurring disease despite adequate testosterone suppression.
* Progression must be evidenced and documented by any of the following parameters:

  * PSA progression defined by a minimum of two rising PSA levels with an interval of greater than or equal to 1 week between each determination
  * Appearance of one or more new lesions consistent with prostate cancer on bone scan
  * New or growing lesions on computed tomography (CT) scan
* Patients must have metastatic disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1(64).
* Patients must have received treatment with prior enzalutamide for two or more cycles and must have had evidence of disease progression while on enzalutamide.
* Patients who have received antiandrogens such as flutamide, bicalutamide, or nilutamide for >6 months immediately before enrollment on this study must be off treatment for 4 weeks (6 weeks for bicalutamide) and demonstrate a continued rise in PSA. Patients on antiandrogens for <6 months must be off medication for 2 weeks.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of enzalutamide and CRLX101 in patients <18 years of age and prostate cancer is not common in children <18 years of age, children are excluded from this study.
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits; for patients with Gilberts syndrome, total bilirubin less than or equal to 3.0 mg/dL
  * hemoglobin greater than or equal to 9g/dL
  * serum albumin greater than or equal to 2.8 g/dL
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT)Serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 times institutional upper limit of normal (<5 times institutional ULN for liver metastases)
  * creatinine within 1.5 times normal institutional limits

OR

--creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.

* Patients must have castrate levels of testosterone (<50 ng/dL [1.74 nmol/L]).
* Patients must have undergone bilateral surgical castration or must continue on gonadotropin-releasing hormone (GnRH) agonists/antagonists for the duration of the study.
* Patients on 5-alpha reductase inhibitors such as finasteride or dutasteride must stop medication at least 28 days prior to study entry.
* The effects of enzalutamide and CRLX101 (formerly IT-101) on the developing human fetus are unknown. For this reason and because androgen receptor antagonists and topoisomerase I inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, all study subjects must agree to use a condom during the study treatment period and for 120 days following the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents. A minimum washout period of 28 days is required prior to the initiation of on study treatment unless the patient is receiving immunotherapy, for which the minimum washout period will be 14 days. This is because Immune-related toxicities are distinct and unlikely to synergize with this protocol therapy, a shorter washout period is reasonable and customary in clinical trials.
* Patients who have been treated with prior secondary hormonal manipulations with proposed investigational rationale for having efficacy against androgen receptor variant 7 (AR-V7) splice variants.

This includes but is not limited to Ralaniten (EPI-002) and AZD5312 (IONIS-AR-2.5Rx). (Note: patients previously treated with abiraterone, orteronel (TAK-700), apalutamide (ARN-509), galeterone, or VT-464 (formerly INO-464) will be eligible for this study. Patients who have received prior chemotherapy will also be eligible for this study).

* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Patients with a recent (within 1 year) history of seizure or any condition that, in the opinion of the investigator, significantly increases seizure risk. Also, current or prior treatment with anti-epileptic medications for the treatment of seizures. Transient ischemic attack within 12 months prior to study enrollment will not be permitted.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to enzalutamide, CRLX101, or other agents used in study.
* Patients with a history within the last 3 years of another invasive malignancy (localized non-melanoma skin and bladder cancers are allowed).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension (systolic blood pressure (SBP)>170/diastolic blood pressure (DBP)>105), or psychiatric illness/social situations within 6 months that would limit compliance with study requirements.
* Patients who have received palliative radiotherapy within 2 weeks of study entry and have not recovered to Grade 1 or baseline from associated toxicities. Note: Patients may receive palliative radiation once enrolled on study. The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) less than or equal to Grade 1 from toxicity due to all prior therapies, including surgery, except alopecia and other non-clinically significant adverse events (AEs).
* Patients who are unable to swallow tablets or have a gastrointestinal disease that could hinder the absorption of enzalutamide
* The use of any herbal products that may lower prostate-specific antigen (PSA) levels (e.g., saw palmetto).
* Patients with microscopic hematuria (defined as >100 red blood cells (RBCs) on urinalysis) or worsening urinary symptoms within 7 days prior to the initiation of study treatment.
* Known human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy are ineligible because of potential pharmacokinetic interactions with study drugs. However, patients with long-standing (>5 years) HIV on antiretroviral therapy >1 month (undetectable HIV viral load and cluster of differentiation 4 (CD4) count > 150 cells/micro L) may be eligible if the Principal Investigator or designee determines no anticipated clinically significant drug-drug

interactions.

INCLUSION OF MINORITIES AND WOMEN:

-Men of all races and ethnic groups are eligible for this trial. Women are excluded as prostate cancer does not exist in this population.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
  All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to the Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- [Derived] Schmidt KT, Karzai F, Bilusic M, Cordes LM, Chau CH, Peer CJ, Wroblewski S, Huitema ADR, Schellens JHM, Gulley JL, Dahut WL, Figg WD, Madan RA. A Single-arm Phase II Study Combining NLG207, a Nanoparticle Camptothecin, with Enzalutamide in Advanced Metastatic Castration-resistant Prostate Cancer Post-Enzalutamide. Oncologist. 2022 Sep 2;27(9):718-e694. doi: 10.1093/oncolo/oyac100. PMID 35640474
- [Derived] Schmidt KT, Chau CH, Strope JD, Huitema ADR, Sissung TM, Price DK, Figg WD. Antitumor Activity of NLG207 (Formerly CRLX101) in Combination with Enzalutamide in Preclinical Prostate Cancer Models. Mol Cancer Ther. 2021 May;20(5):915-924. doi: 10.1158/1535-7163.MCT-20-0228. Epub 2021 Feb 25. PMID 33632874
- [Derived] Schmidt KT, Huitema ADR, Dorlo TPC, Peer CJ, Cordes LM, Sciuto L, Wroblewski S, Pommier Y, Madan RA, Thomas A, Figg WD. Population pharmacokinetic analysis of nanoparticle-bound and free camptothecin after administration of NLG207 in adults with advanced solid tumors. Cancer Chemother Pharmacol. 2020 Oct;86(4):475-486. doi: 10.1007/s00280-020-04134-9. Epub 2020 Sep 8. PMID 32897402
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0096.html

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Lead-In Safety: CRLX101 With Enzalutamide: Lead-in Dosing: CRLX101 (formerly IT-101) 12mg/m^2 every (q) 2 weeks x 2 cycles; CRLX101 15mg/m^2 (q) 2 weeks cycle 3+; enzalutamide 160 mg every day (QD) cycle 1 day 2+
Period: Overall Study
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide | 2/Efficacy: CRLX101 With Enzalutamide
Started | 4 | 0
Completed | 1 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Progressive disease | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.65 (3.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Median Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/ml] — Normal PSA is variable. Higher above the normal range often means more cancer.
  ng/ml | 93.7 [33.7 to 143.0]
Median Prior Lines of Therapy [Median (Full Range); unit: Lines of therapy] — Prior lines of therapy refers to the multiple lines of treatment given to a participant for their disease. First treatment, second treatment, third treatment, and so forth.
  Lines of therapy | 4.5 [4 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Anti-tumor Activity
Description: Anti-tumor activity is >=50% prostate-specific antigen (PSA) decline or stable disease on imaging following 5 months of treatment in participants with progressive metastatic castration resistant prostate cancer (mCRPC) following enzalutamide treatment. Stable disease (SD) is neither sufficient shrinkage to qualify for partial response (at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters) nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study).
Time Frame: 5 months
Measure: Number; unit: percentage of participants
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
percentage of participants
  >=50% prostate-specific antigen (PSA) decline | 25
  Stable Disease | 0

2. Secondary Outcome: Proportion of Participants With a Sustained >30% Decline in Prostate-specific Antigen (PSA)
Description: Proportion of participants with a sustained >30% decline in prostate-specific antigen (PSA) from baseline based on all evaluable participants.
Time Frame: time of sustained >30% decline in prostate-specific antigen (PSA) from baseline, approximately >1 month
Measure: Number; unit: proportion of participants
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
proportion of participants | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the duration of time from the start of treatment to the time of death estimated based on all evaluable participants.
Time Frame: time from the start of treatment to the time of death, up to 17.5 months
Population: 3/4 participants were analyzed because one participant was lost to follow-up.
Measure: Median (Full Range); unit: Months
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 3
Months | 3.9 [3.8 to 17.9]

4. Secondary Outcome: Number of Participants With a Change in Measurable Disease From Baseline as Determined by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Number of participants with a change in measurable disease as determined by RECIST. Complete response (CR) is disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Within 6 months
Measure: Count of Participants; unit: Participants
Groups:
- 1/Lead-In Safety: CRLX101 With Enzalutamide: Lead-in Dosing: CRLX101 12mg/m^2 every (q) 2 weeks x 2 cycles; CRLX101 15mg/m^2 (q) 2 weeks cycle 3+; enzalutamide 160 mg every day (QD) cycle 1 day 2+
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
Participants | 0

5. Secondary Outcome: Number of Participants With a Change in Measurable Disease as Determined by the Prostate Cancer Working Group 3 (PCWG3)
Description: Number of participants with a change in measurable disease as determined by the Prostate Cancer Working Group 3 (PCWG3). PSA values will be captured at each visit and PSA declines and progression (by radiographic evidence or clinical symptoms) will be followed. Radiographic disease progression is considered if a minimum of two new lesions is observed on bone scan. Clinical disease progression is the need for chemotherapy or other change in therapy based on increased cancer related symptoms.
Time Frame: Study end, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
Participants | 0

6. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 26 months and 6 days.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 26 months and 6 days.
Arm/Group | 1/Lead-In Safety: CRLX101 With Enzalutamide
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Lead-In Safety: CRLX101 With Enzalutamide (N=4)
Cystitis noninfective (Renal and urinary disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Lead-In Safety: CRLX101 With Enzalutamide (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Eye disorders - Other, subconjunctival hemorrhage, left eye (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (6)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 1 (5)
Pain (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Dx cough/URI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (2)
White blood cell decreased (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03531827/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT03531827/ICF_001.pdf